CLINICAL TRIAL: NCT05665296
Title: Effect of Cervicothoracic Mobilization on Upper Crossed Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Mohamed Atta El-Kaffas, assistant lecturer of physical therapy-Benha University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003840
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Upper Crossed Syndrome
Keywords: Forward head posture; Rounded Shoulders; Thoracic kyphosis; UCS; Mobilization
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervicothoracic mobilization (Experimental): This group will receive cervicothoracic mobilization with comprehensive corrective exercise
  Interventions: Other: cervicothoracic mobilization; Other: CCE
- control group: comprehensive corrective exercise (CCE). (Active Comparator): This group will receive traditional treatment comprehensive corrective exercise (CCE).
  Interventions: Other: CCE

INTERVENTIONS:
Other: cervicothoracic mobilization — Each participant in study group will receive cervicothoracic mobilization (central PA and transverse Grade III or grade IV) with comprehensive corrective exercise. The duration will eight weeks three sessions per week.
  Arms: cervicothoracic mobilization
Other: CCE — Each participant will receive comprehensive corrective exercise include three phases: Initial phase -Improvement phase and Maintenance phase.
  The initial phase exercises progress in frequency and intensity during this phase, as long as participants are able to demonstrate good quality movement. The initial phase duration is 2 weeks and the exercises will be performed for seven sets of 10-s hold .
  Improvement phase exercises are progressed by considering individual characteristics of each participant and by observing the overload principle and the progression in the number of repetitions of each set during the 4 weeks of the improvement phase. The exercises will be performed from five sets of ten repetitions to six sets of 15 repetitions .
  Maintenance phase exercises:The exercises are the same as in the improvement phase without any progression in intensity and frequency. The maintenance phase duration is 2 weeks

SUMMARY:
PURPOSE: To investigate the effect of cervicothoracic mobilization on Craniovertebral angle (CVA), sagittal shoulder angle (SSA), kyphotic angle and pain intensity level in upper crossed syndrome.

DETAILED DESCRIPTION:
Upper crossed syndrome and its associated neck pain is considered to be the fourth most frequent cause of disability with an annual 30% increase in the rate of prevalence. According to the report on Global burden of diseases (GBD) 2010, neck pain is ranked 21st in terms overall burden of diseases. Musculoskeletal pain in the neck and upper limbs is common; population studies suggest that 6-48% of adults have pain in one of these areas .

Recently, joint mobilization has proven to be effective, and it is now frequently used in clinics .Cervical mobilization combined with thoracic mobilization is recommended as a clinical intervention for neck pain patients with forward head posture ( FHP) rather than cervical mobilization alone. This study has two groups; one will receive cervicothoracic Mobilization + conventional treatment and the second will receive conventional treatment for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-50 years .
2. Participants will included if their CVA less than 48° ( SSA less than 52°) , as above these values are considered normal and thoracic kyphosis (with flexicurve angle more than 45 degrees) .
3. Subjects who have weakness in deep neck flexors, serratus anterior, middle and lower trapezius and rhomboid muscles and tightness in upper trapezius, levator scapulae, scalene, posterior neck and suboccipital muscles, pectoralis major and minor and sternocleidomastoid muscles.
4. Subject complaining of this symptom for more than 3mothes.
5. Marking pain intensity score visual analog scale (VAS) ≥3 in neck and shoulder

Exclusion Criteria:

1. History of surgery or joint diseases of the spine or shoulder.
2. Osteoporosis, or fracture ,cervical instability or any sign those with other contraindications against joint mobilization.
3. Individuals with any cervical condition e.g. radiculopathy, cervical rib, whiplash injury and individuals with any neurological/ condition .
4. History of congenital spinal deformity (congenital scoliosis) .
5. Any malignancy related to soft tissue and joints .
6. Subjects taking analgesics and/or muscle relaxants.
7. pregnancy.
8. Being in weight out of the normal range (18 ≥ BMI ≥ 25).
9. Cognitive impairment and inability to understand the scale.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
change in Craniovertebral angle (CVA) . | before treatment,and after eight weeks of treatment.
  Craniovertebral angle (CVA) will be measured using Computerized photogrammetry is utilized markers, Digital camera and Kinovea software.
change in Sagittal shoulder angle (SSA). | before treatment,and after eight weeks of treatment.
  Sagittal shoulder angle (SSA) will be measured using Computerized photogrammetry is utilized markers, Digital camera and Kinovea software.
change in thoracic kyphosis angle. | before treatment,and after eight weeks of treatment.
  thoracic kyphosis angle will be measured using the flexicurve ruler
change in pain level | before treatment,and after eight weeks of treatment.
  pain severity will be measured using visual analogue scale Each participant will be asked to put a mark on a 10-cm horizontal line that is marked with 'zero' at one end to indicate no pain and marked with'10' at the other end to indicate maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Yamany, professor, Study Chair — Professor of physical therapy, Cairo University

REFERENCES:
- [Background] Seidi F, Bayattork M, Minoonejad H, Andersen LL, Page P. Comprehensive corrective exercise program improves alignment, muscle activation and movement pattern of men with upper crossed syndrome: randomized controlled trial. Sci Rep. 2020 Nov 26;10(1):20688. doi: 10.1038/s41598-020-77571-4. PMID 33244045